CLINICAL TRIAL: NCT07176715
Title: Same-Day Colectomy: is it Safe for Patients?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Eugene Kim, Assistant Clinical Professor, Clinical Series, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003441
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Colorectal; Colectomy; Colectomy Left/Right/Total Under Laparotomy
Keywords: Same Day Colectomy; outpatient Colectomy

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to show that outpatient colectomy is safe and feasible for patients that were rigorously screened preoperatively.
  * The primary outcome of this study is the 30-day rate of readmission to the hospital following same day colectomy.
  * Secondary outcomes include rate of surgical site infection, deep surgical infection, anastomotic leak, bleeding requiring transfusion, postoperative ileus, reoperation, reintervention, acute kidney injury or renal failure, reintubation or need for prolonged ventilation, mortality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Same Day Colectomy (Experimental)
  Interventions: Other: Same-Day Colectomy

INTERVENTIONS:
Other: Same-Day Colectomy — study, they will undergo extensive education during their preoperative visit. Perioperative education includes management of perioperative medications, bowel prep and perioperative antibiotics. Perioperative education will include that of the patient and their designated caregiver.
  Perioperative nursing staff will go over postoperative discharge instructions again. A custom discharge instruction sheet will be made and given to all patients upon discharge. On days 1 and 3 postoperatively, patients will receive a phone call or virtual visit from a member of the research team. Questions will be asked of patients based on a script made. Patients will then be seen in the clinic between postoperative day 5-7.
  Patients' medical record will be followed for six months postoperatively to track emergency department visits, readmissions, and postoperative complications. Postoperative complications will include surgical site infection, deep surgical infection, bleeding requiring transfusion, ana
  Other Names: Outpatient Colectomy

SUMMARY:
This is a prospective cohort study of outcomes of patients undergoing outpatient colorectal surgery at a single institution to study outpatient colectomy as a viable treatment option for a select group of patients requiring colon and rectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Undergoing robotic-assisted right colectomy, sigmoidectomy, or low anterior resection.
* Able to perform greater than 4 metabolic equivalents (METS) without shortness of breath
* Must have a designated adult who can care for them at home postoperatively until their in-person clinic visit
* Access to a cell phone or computer and running water.
* Successfully completed pre-operative and post-operative education
* Medical criteria:
* Well controlled hypertension with systolic blood pressure < 140 controlled by less than two medications which they are compliant with
* Well controlled diabetes on oral agents only with blood glucose level < 180 on daily checks
* Anti-platelet agents including aspirin, clopidogrel, prasugrel, ticagrelor or ticlopidine will be stopped 7 days preoperatively and restarted on postoperative day 1. See exclusion criteria 7 for specific exclusion criteria regarding antiplatelet agents.

Exclusion Criteria:

* Medical criteria:
* Neurocognitive deficits not allowing for adequate preoperative education
* Congestive heart failure with EF < 45%
* Symptomatic aortic stenosis causing heart failure, syncope, dyspnea or angina
* Pulmonary fibrosis or pulmonary hypertension
* COPD or home oxygen use > 2L
* Chronic kidney disease of any stage.
* Lack of a caregiver at home or functionally bed-bound
* Ultralow pelvic resection
* Need for ostomy creation intraoperatively
* Operative time greater than 5 hours as this likely indicates a complex case and dissection necessitating closer monitoring in the hospital
* Conversion to open procedure intraoperatively
* Patients receiving antiplatelet agents such as clopidogrel, prasugrel, ticagrelor or ticlopidine within one year of coronary or carotid stent implantation, TAVR or LAAO placement.
* Patients on therapeutic anticoagulation medications such as warfarin, Eliquis, Xarelto, Enoxaparin
* Current tobacco use
* Patients who were unable to complete preoperative education, do not feel comfortable with care at home, or do not have an available caregiver for the first 7 postoperative days
* Any surgical history that would preclude safe abdominal entry for robotic surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Readmission | 30-Days post-procedure
  The primary outcome of this study is the 30-day rate of readmission to the hospital following same day colectomy

SECONDARY OUTCOMES:
rate of surgical site infection | 30-days Post Procedure
rate of deep surgical infection | 30-days Post Procedure
rate of anastomotic leak | 30-days Post-procedure
rate of bleeding requiring transfusion | 30-Days Post-Procedure
rate of postoperative ileus | 30-Days Post-Procedure
rate of reoperation | 30-Days Post-Procedure
reintervention | 30-Days Post-Procedure
rate of acute kidney injury or renal failure | 30-Days Post-Procedure
rate of reintubation or need for prolonged ventilation | 30-Days Post-Procedure
Rate of mortality | 30-Days Post Procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kim, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourgouin S, Monchal T, Schlienger G, Franck L, Lacroix G, Balandraud P. Eligibility criteria for ambulatory colectomy. J Visc Surg. 2022 Feb;159(1):21-30. doi: 10.1016/j.jviscsurg.2020.11.012. Epub 2020 Dec 19. PMID 33349570
- [Background] Studniarek A, Borsuk DJ, Kochar K, Park JJ, Marecik SJ. Feasibility assessment of outpatient colorectal resections at a tertiary referral center. Int J Colorectal Dis. 2021 Mar;36(3):501-508. doi: 10.1007/s00384-020-03782-w. Epub 2020 Oct 22. PMID 33094353
- [Background] Campbell S, Fichera A, Thomas S, Papaconstantinou H, Essani R. Outpatient colectomy-a dream or reality? Proc (Bayl Univ Med Cent). 2021 Sep 16;35(1):24-27. doi: 10.1080/08998280.2021.1973327. eCollection 2022. PMID 34970026
- [Background] Lee L, Eustache J, Tran-McCaslin M, Basam M, Baldini G, Rudikoff AG, Liberman S, Feldman LS, McLemore EC. North American multicentre evaluation of a same-day discharge protocol for minimally invasive colorectal surgery using mHealth or telephone remote post-discharge monitoring. Surg Endosc. 2022 Dec;36(12):9335-9344. doi: 10.1007/s00464-022-09208-8. Epub 2022 Apr 13. PMID 35419638
- [Background] Gignoux B, Pasquer A, Vulliez A, Lanz T. Outpatient colectomy within an enhanced recovery program. J Visc Surg. 2015 Feb;152(1):11-5. doi: 10.1016/j.jviscsurg.2014.12.004. Epub 2015 Feb 7. PMID 25661787
- [Background] Curfman KR, Poola AS, Blair GE, Kosnik CL, Pille SA, Thilo EL, Hawkins ME, Rashidi L. Ambulatory colectomy: A pilot protocol for same day discharge in minimally invasive colorectal surgery. Am J Surg. 2022 Aug;224(2):757-760. doi: 10.1016/j.amjsurg.2022.04.039. Epub 2022 May 11. PMID 35570059
- [Background] Gignoux B, Gosgnach M, Lanz T, Vulliez A, Blanchet MC, Frering V, Faucheron JL, Chasserant P. Short-term Outcomes of Ambulatory Colectomy for 157 Consecutive Patients. Ann Surg. 2019 Aug;270(2):317-321. doi: 10.1097/SLA.0000000000002800. PMID 29727328
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Papageorge CM, Zhao Q, Foley EF, Harms BA, Heise CP, Carchman EH, Kennedy GD. Short-term outcomes of minimally invasive versus open colectomy for colon cancer. J Surg Res. 2016 Jul;204(1):83-93. doi: 10.1016/j.jss.2016.04.020. Epub 2016 Apr 22. PMID 27451872
- [Background] Miller TE, Thacker JK, White WD, Mantyh C, Migaly J, Jin J, Roche AM, Eisenstein EL, Edwards R, Anstrom KJ, Moon RE, Gan TJ; Enhanced Recovery Study Group. Reduced length of hospital stay in colorectal surgery after implementation of an enhanced recovery protocol. Anesth Analg. 2014 May;118(5):1052-61. doi: 10.1213/ANE.0000000000000206. PMID 24781574